CLINICAL TRIAL: NCT02265146
Title: Association of Lipid Core Plaque With Subsequent Clinical Outcomes: a Collaborative Near-infrared Spectroscopy Study
Brief Title: ORACLE-NIRS: Lipid cORe Plaque Association With CLinical Events: a Near-InfraRed Spectroscopy Study
Acronym: ORACLE-NIRS
Status: Withdrawn | Type: Observational
Why Stopped: 0
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STU 112013-073
Record Dates: First submitted 2014-09-26; First posted 2014-10-15 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Coronary Atherosclerosis
Keywords: Lipid Core Plaques (LCPs); Vulnerable Plaque; Near Infrared Spectroscopy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-center, investigator initiated study that will prospectively examine treatment strategies and outcomes of patients who underwent clinically-indicated Near Infrared Spectroscopy (NIRS). The information collected will be used to determine the frequency of NIRS imaging performed at the participating sites and to examine the clinical outcomes of the NIRS-detected Lipid Core Plaques (LCPs).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone/ will be undergoing NIRS imaging at each of the participating centers.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing clinically-indicated Near Infrared Spectroscopy (NIRS) among various participating centers.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiac events | 1 to 15 years following clinically indicated Near InfraRed Spectroscopy imaging
  The primary endpoint for both hypotheses is the incidence of major adverse cardiac events. Major adverse cardiac events include the following:
  * cardiac death
  * cardiac arrest
  * acute coronary syndrome
  * stent thrombosis, repeat coronary angiography
  * coronary revascularization (either by percutaneous coronary intervention or coronary artery bypass graft surgery).
  * rehospitalization for progressive angina, attributed to a non-culprit lesion secondary to significant fixed, non-reversible (not-spasm related) lesion progression of more than 20% from the baseline study (confirmed by either serial angiography or by necropsy).
  Events will be classified as events occurring at the site of stent implantation and events occurring at previously untreated lesions. Moreover, analyses will be performed on a per patient and per LCP basis.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (5):
- United States (5):
  - North Florida/(South Georgia) VA Health Care System, Gainesville, Florida
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - VA North Texas Health Care System, Dallas, Texas